CLINICAL TRIAL: NCT05511090
Title: Diagnosis and Management of Incidental Pulmonary Nodules: a Prospective Study
Brief Title: Prospective Study to Observe and Manage Progression of Pulmonary Nodules
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Chinese Chronic Respiratory Disease Research Network (Network)
Responsible Party: Sponsor
Other Study IDs: LNs003
Record Dates: First submitted 2022-08-19; First posted 2022-08-22 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: Lung Nodules

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Based on the previous review and research, we would like to further observe the nodule changes in patients with pulmonary nodules. These changes include factors such as the reason for the further enlargement or deterioration of the nodule, time, lifestyle, the patient's region, and hereditary medical history. At the same time, we will further look at the corresponding characteristics of a population that does not change the size and nature of the nodule, including age, gender, and all the factors discussed above. On this basis, we can propose more scientific methods for the treatment and management of pulmonary nodules, and provide a more reliable clinical reference for the clinical treatment of pulmonary nodules.

ELIGIBILITY:
Inclusion Criteria:

LNs patients aged 18 years and older who were previously treated in Guang'anmen hospital.

Exclusion Criteria:

(1) had the LNs removed; (2) LNs less than or equal to 3 mm in size; (3) had not undergone thorax CT; (4) had failed to complete treatment; (5) had incomplete medical records or was lost to follow-up.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: LNs patients aged 18 years and older who were previously treated in Guang'anmen hospital.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Estimated)
Dates: Start 2022-08-30 (Estimated); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in nodule size by CT scan in patients with pulmonary nodules during follow-up. | 6 months
  Changes in nodule size by CT scan in patients with pulmonary nodules during follow-up.